CLINICAL TRIAL: NCT05150470
Title: Evaluation of the Dental Movements Caused by Oral Appliance in Syndrome Sleep Apnea Syndrome(DPOAM)
Brief Title: Evaluation of the Dental Movements Caused by Oral Appliance in Sleep Apnea Syndrome
Acronym: DPOAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Valence (Other)
Collaborators: Claude Bernard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RIPH-CHV-08
Record Dates: First submitted 2021-10-19; First posted 2021-12-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea Syndromes
Keywords: oral appliance; dental movement
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open label (Other): Single Group Assignment
  Interventions: Other: prevention

INTERVENTIONS:
Other: prevention — dental digital fingerprinting
  Other Names: dental digital fingerprinting

SUMMARY:
The DO OAM study is a mono-center, interventional, prospective study carried out in CH VALENCE.

It will estimate the prevalence of dental movements in patients treated by oral Appliance for Sleep Apnea syndrome.

The investigators will used fingerprinting technique by taking multiple photographs of the teeth that allow for the three-dimensional reconstruction of the teeth

this study will provide a better understanding of dental movement caused by oral appliance

DETAILED DESCRIPTION:
oral appliances are indicated for the treatment of Sleep Apnea syndrome. Dentoskeletal effects of oral Appliance are imperfectly assessed.

the investigators want to study dental movements by comparing three-dimensional reconstruction of the teeth and the dental articulation in patients treated for sleep apnea syndrome in our Hospital.

The study consists of an additional acquisition of three-dimensional reconstruction of teeth.

the data previously acquired during the first digital impression according usual practise will be compared to this additional acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of sleep apnea syndrome treated by Oral appliances in CH Valence
* Availability of previous digital impressions required for Oral appliances manufacturing
* Age ≥ 18 years old
* Read, write and understand the French language

Exclusion Criteria:

* Patient under guardianship, deprived of liberty, safeguard of justice
* Refusal to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
dental movement | 1 DAY at inclusion visit only
  dental length rotation (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Buiret, Principal Investigator — CH VALENCE
Locations (1):
- Ch Valence, Valence, France

IPD SHARING:
Plan to Share IPD: No